CLINICAL TRIAL: NCT00676936
Title: Corticosteroids for Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OPI 07-005; 2007-005617-19 (EudraCT Number)
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Cancer; Pain
Keywords: Cancer; pain; corticosteroids; palliative; supportive care; Cancer patients with pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylprednisolone (Experimental): Methylprednisolone 16 mg twice daily
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): Placebo capsules twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Custom made capsules, Methylprednisolone 16 mg twice daily, intervention period 7 days.
  Other Names: Medrol (TM)
  Arms: Methylprednisolone
Drug: Placebo — Custom made capsules, Lactose, administered twice daily, intervention period 7 days
  Arms: Placebo

SUMMARY:
Study hypothesis: corticosteroids are effective for pain in cancer patients. We will perform a double-blind, randomized, placebo-controlled multicentre trial evaluating the effect of Methylprednisolone 16 mg twice daily in cancer patients with pain (average pain last 24 hrs NRS > 4 (Numerical rating scale, 0 No pain, 10 worst pain).

DETAILED DESCRIPTION:
Patients are required to use strong opioids before entering the study. Weak opioids are allowed if patients have short acting strong opioids as rescue-medication. The scheduled opioids shall be stable last 48 hours before entering the study and will be kept stable during the study period. Patients may use as much short acting rescue-medication as they require. No other analgesic medication should be started during the study period.

The study is a multicentre trial. Patients will be randomized according to 1. study centre (No 1-5) and 2. pain mechanism: skeletal metastases (yes/no).

Patients are evaluated Day 0 and Day 7 by palliative care physician. Patients will be contacted by phone Day 1-6 and will fill in questionnaire regarding symptoms and analgesic usage. Patients will be contacted Day 14 and 21 to fill in questionnaires regarding symptoms, quality of life and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Verified malignant disease
* Receiving a scheduled strong or weak opioid
* Insufficient pain control: Average pain last 24 h: ≥ 4 (NRS 0-10)
* Given informed consent according to the ethical guidelines
* Able to complete planned assessment schedules
* ≥ 18 years of age
* Life expectancy > 1 month

Exclusion Criteria:

* Excruciating pain (average pain ≥ 8) (These patients should be considered as emergency patients. Patients may be eligible for the study after stabilization)
* Dose adjustment in scheduled opioid medication last 48 hours
* Concurrent medication with NSAIDs (Patients are eligible for the study one week after NSAIDs are discontinued)
* Receiving radiotherapy within 4 weeks before entering the study or planned within the study period
* Started systemic treatment (chemotherapy, hormone therapy or bisphosphonates) within 4 weeks before entering the study Patients who have received chemotherapy for more than 4 weeks are eligible for the study if it is more than 7 days since receiving the last dose and they are not having the next dose within the study period
* Manifest spinal cord compression or in need of bone surgery
* Severe cognitive impairment
* Previously on steroids during the last 4 weeks
* Diabetes mellitus
* Known peptic ulcer disease
* Systemic fungal disease, patients vaccinated with viable viruses, and patients with known allergies to the study medication (MethylPrednisolone)
* Female patients who are pregnant or lactating.
* Women of reproductive potential not willing or unable to employ an effective method of contraception (be sterilized, using IUD or oral contraception)
* Patients using following medication: cyclosporin, erythromycin, phenobarbital, phenytoin, carbamazepin, ketoconazole, methotrexate, ciclofosfamide, rifampicin, aprepitant and diltiazem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
pain intensity at Day 7 | 7 days
  change of pain intensity at Day 7, measured by "average pain for the last 24 hours" (NRS 0-10).

SECONDARY OUTCOMES:
fatigue | 7 days
  change of fatigue measured by EORTC QLQ30 and ESAS
appetite | 7 days
  change of appetite measured by EORTC QLQ30 and ESAS
Overall effect satisfaction | 7 days
  Overall effect measured by a global satisfaction-question ("How is your overall benefit from the medication?" NRS: 0= No important benefit 10=very important benefit).
sleep quality | 7 days
  change of sleep quality measured by Pittsburgh Sleep Quality Index
analgesic usage | 7 days
  change of analgesic usage measured by morphine equivalents.
Pain now and average pain last 24 hrs | 7 days
  Pain now and average pain last 24 hours measured by daily NRS (Numeric rating scale)(ESAS)

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD PhD prof, Study Director — Norwegian University of Science and Technology
Locations (6):
- Norway (6):
  - Haraldsplass Diakonale sykehus, Bergen
  - Sykehuset Buskerud HF, Drammen
  - Sørlandet Sykehus HF, Kristiansand
  - Oslo Universitetssykehus, Ulleval, Oslo
  - Sykehuset Telemark HF, Skien
  - St Olavs Hospital HF, Trondheim

REFERENCES:
- [Result] Paulsen O, Klepstad P, Rosland JH, Aass N, Albert E, Fayers P, Kaasa S. Efficacy of methylprednisolone on pain, fatigue, and appetite loss in patients with advanced cancer using opioids: a randomized, placebo-controlled, double-blind trial. J Clin Oncol. 2014 Oct 10;32(29):3221-8. doi: 10.1200/JCO.2013.54.3926. Epub 2014 Jul 7. PMID 25002731
- [Result] Jakobsen G, Engstrom M, Hjermstad MJ, Rosland JH, Aass N, Albert E, Kaasa S, Fayers P, Klepstad P, Paulsen O. The short-term impact of methylprednisolone on patient-reported sleep in patients with advanced cancer in a randomized, placebo-controlled, double-blind trial. Support Care Cancer. 2021 Apr;29(4):2047-2055. doi: 10.1007/s00520-020-05693-6. Epub 2020 Aug 27. PMID 32856209